CLINICAL TRIAL: NCT04087005
Title: Efficacy and Safety of JHG002(Hominis Placenta, 紫河車) Therapy for Chronic Temporomandibular Joint Dysfunction: A Multicenter Randomized Controlled Trial)
Brief Title: Efficacy and Safety of JHG002 for Chronic Temporomandibular Joint Dysfunction: A Multicenter Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2017-04
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hominis placental pharmacopuncture (Experimental): The Hominis placental pharmacopuncture group will receive 10 sessions of Hominis placental pharmacopuncture at 2 sessions/week for 5 weeks. A trained doctor of Korean medicine with at least 2 years clinical experience will administer JHG002 pharmacopuncture with a disposable syringe (0.5ml) directly into the designated sites, using a standardized method.
  Interventions: Other: hominis placental pharmacopuncture
- Transcutaneous electrical nerve stimulation (Active Comparator): The control group will receive 2 sessions/week of TENS for 5 weeks. A high-frequency, low-intensity stimulus of 50-100Hz and up to 15mA will be used, such that the patients feel a current but do not feel pain. At each treatment visit, a physiotherapist will administer the treatment to the bilateral temporomandibular joint for 15 minutes. Both centres will use the same TENS device-a BioTron-DX (D.M.C, Osan, South Korea).
  Interventions: Other: hominis placental pharmacopuncture

INTERVENTIONS:
Other: hominis placental pharmacopuncture — Hominis placental pharmacopuncture is human placental extract, which has been used in traditional Korean medicine to treat chronic diseases, including frailty, cough, anorexia, and fatigue, by enhancing the body's resistance.

SUMMARY:
This study is a 2-arm parallel, assessor blinded, multi-centre, randomised controlled trial.

DETAILED DESCRIPTION:
From 2 hospitals of Korean medicine, we will enrol 82 chronic TMD patients in Axis 1, Group Ⅰ according to RDC/TMD diagnostic criteria, and randomly allocate 41 patients each to an HPP group and a physical therapy (PT) group. Treatment will be administered in 10 rounds, after which there will be 4 follow-up visits (6, 9, 13, and 25 weeks from baseline). The primary end point is 6 weeks after baseline, and the primary outcome is the difference in Visual analogue scale (VAS) score for temporomandibular pain between baseline and Week 6. Secondary outcomes will be Numeric rating scale (NRS) scores for temporomandibular pain and discomfort, temporomandibular joint range of motion, Korean version of Beck's Depression Index-Ⅱ(K-BDI-II), Jaw Functional Limitation Scale (JFLS), Patien Global Impression of Change(PGIC), and quality of life. Using data on adverse events and cost-effectiveness in the two groups, we will perform a safety assessment and a cost-effectiveness analysis (economic assessment).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral or bilateral TMJ pain
2. Patients with VAS≥40mm for the area showing TMJ pain (for patients with bilateral pain, the side with worse pain)
3. Patients complaining of persistent of sporadic TMJ pain for at least 3 months
4. Patients diagnosed as myofascial TMD (Axis I: Group 1) based on the RDC/TMD diagnostic criteria[5]
5. Patients aged 19-70 years on the date they sign the consent form
6. Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

1. Patients whose current pain episode developed or worsened because of a road traffic accident or traumatic injury
2. Patients diagnosed in Group 2 or 3 of Axis I based on the RDC/TMD diagnostic criteria
3. Patients who have undergone surgery related to the TMJ
4. Patients with other chronic disease that could interfere with interpretation of the treatment effects or outcomes (e.g., rheumatoid arthritis, neoplastic disease, stroke, or myocardial infarction)
5. Patients currently taking steroids, immunosuppressants, psychiatric drugs, or other drugs that could affect the study results
6. Patients who have received HPP within the last month, or who have taken drugs that could affect pain, such as NSAIDs, within the last week
7. Pregnant or breastfeeding women
8. Patients who have finished participation in another clinical trial within the last month, who participated in another trial within 6 months of selection, or who are planning to participate in another clinical trial during the follow-up period
9. Patients with a history of hypersensitivity after HPP
10. Diabetic patients with uncontrolled blood glucose (fasting blood glucose ≥180mg/dl)
11. Patients with AST (GOT) or ALT (GPT) at least 2 times the normal range at the testing centre
12. Patients with creatinine at least 2 times the normal range at the testing centre
13. Patients suspected to have organic disease
14. Patients with cardiac, hepatic, renal, or other serious complications
15. Patients with psychogenic disease
16. Patients who are unable to receive pharmacopuncture due to e.g., inflammation or a wound at the relevant acupoints
17. Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
The difference in visual analogue scale (VAS) of temporomandibular pain | Week 6
  The primary outcome is the difference in VAS for TMJ pain between baseline and the primary end point (Week 6). VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of TMJ pain and discomfort | Week 6
  The extent of TMJ pain and discomfort in the last week will be assessed using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their TMJ pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
TMJ range of motion | Week 6
  A Therabite Range of Motion Ruler will be used to measure the range of TMJ mouth opening and excursive movement; the measurement method will follow the guidelines provided by the International RDC/TMD Consortium.
Korean version of Beck's Depression Index-Ⅱ (K-BDI-Ⅱ) | Week 6
  The BDI-Ⅱ is an index for diagnosing depression, consisting of 21 questions related to sadness, guilt, suicidal ideation, and loss of interest. In this study, we will use the K-BDI-II, which has been demonstrated to be valid and reliable by a Korean research group.
Jaw Functional Limitation Scale (JFLS) | Week 6
  The JFLS is an index assessing jaw function (mastication, mobility, and emotional and verbal expression) in the last month. The instrument consists of 20 questions, and each question is scored 0-10, where 0 points is 'no impairment' and 10 points is 'very severe impairment'. In this study, we will use the official Korean version of the 20-question JFLS, which has been demonstrated to be reliable.
Patient Global Impression of Change (PGIC) | Week 6
  The PGIC is an index that assesses improvements in functional limitation caused by TMD in 7 grades. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.
The five level version of EuroQol-5 Dimension (EQ-5D-5L) | Week 6
  The EQ-5D-5L is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D-5L consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, we will use the Korean version of the EQ-5D-5L, which has been demonstrated to be valid.
SF-12 | Week 6
  The SF-12 is a shortened version of the Short Form-36 Health Survey (SF-36), which is a widely used instrument to assess health-related quality of life. The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life. In this study, we will use the Korean version of the SF-12, which has been demonstrated to be reliable and valid.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (2):
- South Korea (2):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Kyung Hee University Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim D, Kim ES, Kim KW, Cho JH, Lee YJ, Ha IH. Cost-Effectiveness of Hominis Placenta Therapy for Chronic Temporomandibular Disorder: An Economic Evaluation Alongside a Pragmatic Randomised Controlled Trial. J Oral Rehabil. 2025 Jun;52(6):807-816. doi: 10.1111/joor.13932. Epub 2025 Feb 3. PMID 39895393
- [Derived] Park KS, Kim ES, Kim KW, Cho JH, Lee YJ, Lee J, Ha IH. Effectiveness and safety of hominis placental pharmacopuncture for chronic temporomandibular disorder: A multi-center randomized controlled trial. Integr Med Res. 2024 Jun;13(2):101044. doi: 10.1016/j.imr.2024.101044. Epub 2024 Apr 20. PMID 38779539
- [Derived] Kim J, Park KS, Lee YJ, Kim KW, Cho JH, Ha IH. Efficacy, safety, and economic assessment of hominis placental pharmacopuncture for chronic temporomandibular disorder: a protocol for a multicentre randomised controlled trial. Trials. 2020 Jun 15;21(1):525. doi: 10.1186/s13063-020-04442-8. PMID 32539850